CLINICAL TRIAL: NCT01733550
Title: ICare Self-tonometry - A Head-to-head Comparison to the Gold Standard Goldmann Tonometer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: s54640
Record Dates: First submitted 2012-10-31; First posted 2012-11-27 (Estimated); Last update posted 2012-11-28 (Estimated); Status verified 2012-09

CONDITIONS: Glaucoma
Keywords: Intraocular Pressure; Tonometry, Ocular; iCare
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Glaucoma patients: Intraocular pressure is measured by Home iCare performed by the study nurse, by the patient it self and by Goldmann applanation tonometry.
  Interventions: Device: Home iCare (study nurse); Device: goldmann applanation tonometry; Device: home iCare (by patient)

INTERVENTIONS:
Device: Home iCare (study nurse) — the intraocular pressure is measured by iCare performed by the study nurse
Device: goldmann applanation tonometry — the intraocular pressure is measured by goldmann applanation tonometry
Device: home iCare (by patient) — the intraocular pressure is measured by the iCare performed by the patient him self

SUMMARY:
The purpose of this study is to compare glaucoma patients' own I Care measurements by the standard Goldmann applanation tonometer intraocular pressure (IOP) measurements.

DETAILED DESCRIPTION:
not necessary

ELIGIBILITY:
Inclusion Criteria:

* Ocular hypertension (OHT):with/without glaucoma drugs
* Primary open angle glaucoma (POAG)- high pressure: Diagnosis based on optic nerve head rim loss and/or visual field defects and intraocular pressure (IOP) >21 mmHg.
* Primary open angle glaucoma, normal pressure: cfr high pressure but intraocular pressure ≤ 21 mmHg
* Exfoliative Glaucoma (PEX): Diagnosis based on optic nerve head rim loss and/or visual field defects and intraocular pressure (IOP) >21 mmHg, with exfoliation material in the anterior segment.
* Pigmentary Glaucoma (PDG): Diagnosis based on optic nerve head rim loss and/or visual field defects and intraocular pressure (IOP) >21 mmHg, with Krukenberg's spindle and/or pigment dispersed on the trabecular meshwork.

Exclusion Criteria:

* Age <18 years
* Other glaucoma types
* Corneal pathology (edema, dystrophia, corneal transplantation, severe keratoconus, permanent contact lens wear, recurrent corneal erosion)
* Severe arthritis (unable to handle home i care device)
* Lack of comprehension
* Intra ocular surgery and laser treatment during the last 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Glaucoma patients who are admitted to the hospital for repeated eye pressure measurements learn how to handle the home i care during their stay.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2012-11; Primary Completion 2013-04 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
Intra-ocular pressure with Home ICare and Goldmann Applanation Tonometer. | immediate comparison, no time frame required
  Patients eye pressure measurement with both devices.
  1. Home ICare measurement by study nurse compared to Home ICare by patient compared to Goldmann ATO by study nurse (once for every patient)
  2. 4 times daily: measurement Goldmann ATO (by resident in ophthalmology) and home Icare (by patient)on same moment

SECONDARY OUTCOMES:
Patient Comfort | 1 day hospitalisation
  The comfort of the patients will be checked with both methods (home iCare and goldmann applanation tonometry) and look if the patient has a preference for one of them. Pain and discomfort were scaled from 0 to 5 (0 = none,1-2 = slight, 3-4 = moderate, 5 = severe) for both tonometers, and patients were asked which tonometer they preferred.

CONTACTS AND LOCATIONS:
Overall Officials: Ingeborg Stalmans, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- UZLeuven, Leuven, Belgium